CLINICAL TRIAL: NCT07159971
Title: Family-based Intervention Model to Prevent Childhood Obesity Among Schoolage Children in Sonora, Mexico.
Brief Title: Family-Based Nutrition Intervention to Prevent Overweight and Obesity in School-Age Children.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Claudia Teresa Tovar Palacio (Other)
Collaborators: Fundación Gonzalo Río Arronte (Unknown); Instituto Nacional de Medicina Genomica (Other Government); University of Illinois at Urbana-Champaign (Other); Universidad Nacional Autonoma de Mexico (Other)
Responsible Party: Sponsor-Investigator, Claudia Teresa Tovar Palacio, Dr., Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Organization: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 3738
Record Dates: First submitted 2025-07-07; First posted 2025-09-08 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-06

CONDITIONS: Overweight and/or Obesity; Children - Malnutrition; Preventing Malnutrition
Keywords: Obesity; Children; mHealth; Intervention; Family-base
MeSH Terms: conditions — Child Nutrition Disorders; Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- School B (Experimental): Nutritional therapy supported by a mobile application. The app integrates a multimodal approach (educational content, interactive tools, and gamification) to promote healthy eating, featuring parent-child dyad-focused resources such as recipe tutorials with family-specific adaptations.
  Interventions: Device: School B
- School A. (Active Comparator): Nutritional therapy will be delivered through a mobile application that will integrate a multimodal approach, including educational content, interactive tools, and gamification, to promote healthy eating. The application will incorporate parent-child dyad-focused resources, such as recipe tutorials adapted to specific family needs.
  Interventions: Other: Control

INTERVENTIONS:
Device: School B — Nutritional therapy supported by a mobile application.
  Arms: School B
Other: Control — Conventional nutritional treatment.
  Arms: School A.

SUMMARY:
This proposal aims to enhance the well being of schoolchildren and their families through a mobile application and multidisciplinary intervention model grounded in authoritative parenting principles and social cognitive theory.

DETAILED DESCRIPTION:
Childhood is recognized as a critical period of metabolic sensitivity, during which excess adiposity increases the likelihood of developing metabolic abnormalities in adulthood by approximately 70%, including hypertension, dyslipidemia, insulin resistance, hyperuricemia, and non-alcoholic fatty liver disease. In Mexico, overweight and obesity affect 35.5% of school-aged children, inevitably contributing to the growing prevalence of non-communicable chronic diseases. Data from ENSANUT 2018 place Sonora among the five states with the highest rates of obesity, with 22.2% of adolescents aged 12-19 years classified as obese. This epidemiological context highlights the pressing need for innovative strategies to promote prevention and early risk detection during childhood.

Evidence indicates that mobile health (mHealth) applications may effectively reduce body weight and prevent fat accumulation. Nevertheless, only a limited number of studies have applied mHealth interventions to prevent pediatric adiposity or to foster behavioral changes in comparison with conventional nutritional approaches. The proposed model incorporates a communication strategy designed to monitor participant needs, offer engagement incentives, and promote adherence to the study protocol.

The primary research question addresses whether a family-focused intervention can effectively improve eating patterns and food-related behaviors among students enrolled at "La Caridad" Educational Center in Nacozari de García, Sonora.

ELIGIBILITY:
Inclusion Criteria:

* Families of children between 5 and 9 years old.
* Children without any medical or nutritional treatment for obesity.
* Children classified as normal weight, overweight, or obese based on WHO (Z-score: height for age and BMI for age).
* Offspring of mothers aged between 18 and 45 years at delivery.
* Term infants from normoevolutive pregnancies without maternal comorbidities.
* Families who have a cell phone with internet access and an installed camera.

Exclusion Criteria:

* Children who are currently suffering from a pathology that requires medication or special treatment
* Mothers/Fathers/Guardians who are currently suffering from a pathology that requires medication or special treatment.
* Children who have a physical/mental impairment to perform physical activities.
* Children from surrogate mothers who have presented at least 2 of the 11 DSM-5 criteria for substance use disorder (alcohol, tobacco, cannabis, or other illegal drugs) before or during the participating child's gestation.
* Children from multiple pregnancies.
* Parents who do not own a smartphone compatible with the app will be excluded from this study (i.e., version 5.0 or higher for Android).

Ages: 5 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2025-06-30 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Dietary behavior | Six months
  The Children's Eating Behavior Questionnaire (CEBQ) will be administered. The responses will be scored and interpreted using standardized scales, yielding two main dimensions: overeating-related behaviors (where higher scores indicate increased risk of obesity) and undereating-related behaviors (where higher scores suggest risk of underweight or feeding difficulties). Each dimension is further divided into four subscales, allowing for a more detailed characterization of eating behavior patterns.
Body index mass | Six months
  Measured in Kg/m2
Age | Six months
  Years lived reported by parents through medical records
Feeding practices | Six months
  Comprehensive Feeding Practices Questionnaire (CFPQ). The CFPQ evaluates parental feeding behaviors across two primary domains, each comprising six subscales. The first domain encompasses health-promoting feeding practices (e.g., modeling, monitoring), while the second includes negative or problematic feeding practices (e.g., use of food as a reward, restrictive practices). Higher scores in health-promoting practices are positively associated with healthier dietary patterns in children. In contrast, higher scores in negative practices are linked to an increased risk of pediatric obesity and disordered eating behaviors.
Body weight | Six months
  The total body weight (kg) observed in the intervention group versus the control group.
Phisical activity | Six months
  This questionnaire assesses children's average physical activity (expressed in MET-minutes per week) and sedentary time (in hours/day) across weekdays
Height | Six months
  Mean values of anthropometric measurements obtained using a stadiometer, expressed in centimeters.
Fat mass | Six months
  Children's fat mass, as determined by bioelectrical impedance analysis, will be expressed as a percentage (%).
Fat-free mass | Six months
  Children's fat-free mass, as determined by bioelectrical impedance analysis, will be expressed as a percentage (%).
Glucose | Six months
  Change in glucose concentration will be determined by measuring capillary blood glucose levels (mg/dL)
Triacylglycerides | Six months
  Changes in triacylglycerol concentration will be determined by measuring capillary blood triacylglycerol levels (mg/dL)
Total cholesterol | Six months
  Changes in total cholesterol concentration will be determined by measuring capillary blood cholesterol levels (mg/dL).
HDL-Cholesterol | Six months
  Changes in HDL-cholesterol concentration will be determined by measuring capillary blood HDL-cholesterol levels (mg/dL).
LDL-cholesterol | Six months
  Changes in LDL-cholesterol concentration will be determined by measuring capillary blood LDL-cholesterol levels.
Parenting practices | Six months
  The Short Parenting Practices Questionnaire is designed to identify and classify parenting styles based on two primary dimensions: warmth (affection) and control (discipline).
  In its abbreviated version, the questionnaire asks parents/caregivers to report on items that explore:
  Authoritative practices: characterized by high warmth and high control, reflected in behaviors such as providing explanations, setting clear rules, showing affection, and promoting autonomy within appropriate limits.
  Authoritarian practices: characterized by low warmth and high control, reflected in behaviors such as rigid discipline, imposing rules without dialogue, and lower expression of affection.
  In general, the questionnaire requires self-reported responses regarding the frequency with which parents engage in specific behaviors or strategies in everyday life. These responses are then grouped into the two empirically validated categories.
Dietary patterns | Six month
  Using data collected from a food frequency questionnaire (FFQ) and a 24-hour dietary recall will be evaluated for dietary patterns

SECONDARY OUTCOMES:
Z-Score | Six months
  Change in Z-score scale:
  1. - BMI for age: ≤-3SD is equivalent to severe thinness, ≤-2 is equivalent to thinness, ≥+2 is equivalent to obesity and ≥+1 is equivalent to overweight
  2. - Height for age: ≥ -1 is equivalent to normal, ≥-2 to ≤ -1 is equivalent to moderately stunted and ≤ -2 is equivalent to severely stunted

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Tovar-Palacio, Ph.D., Principal Investigator — Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Locations (1):
- "El globo" and "Servicios de Salud Lomas Altas", México, Sonora, Mexico

IPD SHARING:
Plan to Share IPD: No